CLINICAL TRIAL: NCT03813407
Title: An Open-label Study to Assess Safety and Efficacy of SZC in Paediatric Patients With Hyperkalaemia
Acronym: PEDZ-K
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9481C00001; 2023-508455-38-00 (Registry Identifier: CTIS (EU)); 2018-001331-48 (EudraCT Number)
Record Dates: First submitted 2018-11-22; First posted 2019-01-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Hyperkalaemia
Keywords: sodium zirconium cyclosilicate; Hyperkalaemia in children
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate; Streptozocin

STUDY DESIGN:
Intervention Model Description: Treatment includes 3phases:CP,MP,LTMP Eligible participants with hyperkalaemia will enter CP receiving fixed dose of SZC three times daily(TID) for up to 3days until normokalaemia.Within each cohort 2 to<18 years,initial participants will be allocated to dose level (DL)5g TID.After recommendation of higher DLs by iDMC,subsequent participants may be allocated in the CP to 10g TID and potentially 15g TID.Participants in 0 to<2 years cohort will be assigned to the same DL decided based on data from older cohorts.Those who achieve normokalaemia in the CP will enter a 28-day MP,which starts with once daily administration of the dose received TID in the CP.During MP,the Investigator is able to titrate the dose up or down in the range 2.5gto15g body weight equivalent to maintain normokalaemia.For participants who,at the end of MP,are normokalaemic/hyperkalaemic without being on maximum dose,the MP is followed by option to continue in an LTMP where the same titration regimen is used as in MP.
Masking Description: All phases in the study are open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Arm ( Sodium Zirconium Cyclosilicate SZC) (Experimental): Dosage formulation: 5 g sachets 2.5 g sachets 0.25 g sprinkle capsules 0.125 g sprinkle capsules (can be manufactured to support participants <2 years of age) Route of administration: Oral Dosing instructions: SZC is provided as a powder. At the time of dosing SZC is mixed with a quantity of water or sprinkled onto semi-solid food (eg, milk, baby food, yogurt, or ice cream) within an hour of drug administration. Packaging and labelling: Study treatment will be provided in sachets packed in cartons or sprinkle capsules in high density polyethylene bottles, as appropriate for the dose. Each carton of sachets, individual sachets, and bottle of capsules will be labelled in accordance with Good Manufacturing Practice Annex 13 and per country regulatory requirement. Participant-specific dosing cards (diary) will be provided.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (SZC) Reduced Dose Level; Drug: Sodium Zirconium Cyclosilicate (SZC) Dose Level 1 (DL1); Drug: Sodium Zirconium Cyclosilicate (SZC) Dose Level 2 (DL2); Drug: Sodium Zirconium Cyclosilicate (SZC) Dose Level 3 (DL3); Drug: Sodium Zirconium Cyclosilicate (SZC) Dose During 28 Day Maintenance Phase

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (SZC) Reduced Dose Level — Sodium Zirconium Cyclosilicate (SZC) Dose: Paediatric dose based on body weight equivalent to an adult 2.5 g
Drug: Sodium Zirconium Cyclosilicate (SZC) Dose Level 1 (DL1) — Sodium Zirconium Cyclosilicate (SZC)Paediatric dose based on body weight equivalent to an adult 5 g
Drug: Sodium Zirconium Cyclosilicate (SZC) Dose Level 2 (DL2) — Sodium Zirconium Cyclosilicate (SZC) Paediatric dose based on body weight equivalent to an adult 10 g
Drug: Sodium Zirconium Cyclosilicate (SZC) Dose Level 3 (DL3) — Sodium Zirconium Cyclosilicate (SZC) Paediatric dose based on body weight equivalent to an adult 15 g
Drug: Sodium Zirconium Cyclosilicate (SZC) Dose During 28 Day Maintenance Phase — A 28-day period during which SZC is administered orally once daily (QD) to maintain normokalaemia. A dose titration regimen starting with QD administration of the dose of SZC the participants received TID in the CP will be studied in the MP and continued in the LTMP. The maximum dose that can be used is the calculated body weight equivalent to the 15 g adult dose

SUMMARY:
Sodium zirconium cyclosilicate has been shown to be effective and safe in adults for the treatment of hyperkalaemia, and therefore it is expected to be beneficial in children. This study will evaluate the efficacy, safety and tolerability of sodium zirconium cyclosilicate for the treatment of hyperkalaemia in children <18 years of age. Approximately 140 participants will enter CP at approximately 46 sites in locations including but not limited to Europe and North America for this study. Treatment will include 3 phases: the CP, MP, and LTMP. Enrolment will start in 2 cohorts, ages 6 to < 12 years and 12 to < 18 years. After review of accumulated data, the independent Data Monitoring Committee (iDMC) will recommend whether to open enrolment in the ages 2 to < 6 years cohort and later in the ages 0 to < 2 years cohort. All eligible participants with hyperkalaemia will enter an open-label Correction Phase (CP) receiving a fixed dose of SZC three times daily (TID) for up to 3 days until normokalaemia is achieved. Within each age cohorts 2 to < 18 years, initial participants will be allocated to the dose level (DL) based on body weight equivalent to an adult 5 g TID. After recommendation of higher DLs by the iDMC, subsequent participants may be allocated in the CP to on body weight equivalent to an adult 10 g TID and then potentially on body weight equivalent to an adult 15 g TID. All participants in the ages 0 to < 2 years cohort will be assigned to the same DL which will be decided based on data from older age cohorts. Participants who successfully achieve normokalaemia in the CP will enter a 28-day open-label Maintenance Phase (MP), which will be initiated with once daily administration of the dose received TID in the CP. During MP, the Investigator is able to titrate the dose up or down in the range 2.5 g to 15 g body weight equivalent to maintain normokalaemia. For participants who, at the end of MP, are normokalaemic or hyperkalaemic without being on maximum dose, the MP is followed by the option to continue the study in a long term maintenance phase (LTMP) where the same titration regimen is used as in MP

DETAILED DESCRIPTION:
Protocol title: An open-label study to assess safety and efficacy of SZC in paediatric patients with hyperkalaemia

Rationale: Sodium zirconium cyclosilicate has been shown to be effective and safe in adults for the treatment of hyperkalaemia, and therefore it is expected to be beneficial in children. This study will evaluate the efficacy, safety and tolerability of sodium zirconium cyclosilicate for the treatment of hyperkalaemia in children <18 years of age

Primary Objective: Correction phase (CP) primary objective:

1. To evaluate the ability to achieve normokalaemia during the CP when initiating treatment with SZC of different dose levels (DLs) in children with hyperkalaemia 28-day Maintenance Phase (MP) primary objective:
2. To evaluate the ability to maintain normokalaemia during the MP when continuing SZC treatment in children achieving normokalaemia

   Secondary Objectives: All phases secondary objective:
3. To evaluate the change in S-K+ in children treated with SZC

   MP secondary objectives:
4. To evaluate change in serum aldosterone levels in children treated with SZC during the MP
5. To evaluate change in serum electrolytes (including bicarbonate), spot urinary pH and urinary electrolytes levels in children treated with SZC during the MP

   Long-term MP (LTMP) secondary objectives:
6. To evaluate the ability of maintaining normokalaemia in children treated with SZC during the LTMP

   Safety Objective:
7. To evaluate the safety and tolerability of SZC in the 3 phases (CP, MP, and LTMP)

   Tertiary/Exploratory:
8. To evaluate the acceptability and palatability of SZC through the study

Overall design: This is a Phase 3, international, multi-centre, open-label study assessing different doses of SZC. The population to be studied is hyperkalaemic children < 18 years. Dosing will mirror the regimen approved for adults using body weight equivalent doses. Enrolment will start in 2 cohorts, ages 6 to < 12 years and 12 to < 18 years. After review of accumulated data, the independent Data Monitoring Committee (iDMC) will recommend whether to open enrolment in the ages 2 to < 6 years cohort and later in the ages 0 to < 2 years cohort.

The study will be conducted in approximately 11 countries and 46 sites. All eligible participants with hyperkalaemia will enter an open-label Correction Phase (CP) receiving a fixed dose of SZC three times daily (TID) for up to 3 days until normokalaemia is achieved. Within each age cohorts 2 to < 18 years, initial participants will be allocated to the dose level (DL) based on body weight equivalent to an adult 5 g TID. After recommendation of higher DLs by the iDMC, subsequent participants may be allocated in the CP to on body weight equivalent to an adult 10 g TID and then potentially on body weight equivalent to an adult 15 g TID. All participants in the ages 0 to < 2 years cohort will be assigned to the same DL which will be decided based on data from older age cohorts.

Participants who successfully achieve normokalaemia in the CP will enter a 28-day open-label Maintenance Phase (MP), which will be initiated with once daily administration of the dose received TID in the CP. During MP, the Investigator is able to titrate the dose up or down in the range 2.5 g to 15 g body weight equivalent to maintain normokalaemia. The MP is followed by the option for participants to continue the study in a long-term maintenance phase (LTMP) where the same titration regimen is used as in MP, but with monthly visits.

Study period: Estimated date of first participant enter the CP Q4 2018. Estimated date of last participant completed 27 December 2024.

Number of participants: This study aims to enter into CP a total of approximately 140 participants with hyperkalaemia. Of these, approximately 85 participants are expected to have moderate to severe hyperkalaemia. Enrolment will continue until at least 54 participants with moderate to severe hyperkalaemia have entered the MP and 45 participants with moderate to severe hyperkalaemia have completed the MP. A maximum of 55 participants with mild hyperkalaemia will enter the CP. In addition, there are minimum requirements for participants in each age cohort

Duration: Study duration is approximately 28 weeks including up to 3 days of correction treatment, followed by maintenance treatment for 28 days, a LTMP for up to 22 weeks, and a safety follow-up visit 1 week after the last dose.

Treatments and treatment duration:

Treatment will include 3 phases: the CP, MP, and LTMP. All age cohorts are eligible to participate in all phases of the study. The 3 treatment phases are specified below:

Correction phase (CP): All eligible participants with hyperkalaemia will enter an open-label Correction Phase (CP) receiving a fixed dose of SZC three times daily (TID) for up to 3 days until normokalaemia is achieved. Within each age cohorts 2 to < 18 years, initial participants will be allocated to the dose level (DL) 5 g TID. After recommendation of higher DLs by the iDMC, subsequent participants may be allocated in the CP to 10 g TID and then potentially 15 g TID. All participants in the ages 0 to < 2 years cohort will be assigned to the same DL which will be decided based on data from older age cohorts.

Maintenance phase (MP): Participants who successfully achieve normokalaemia in the CP will enter a 28-day open-label Maintenance Phase (MP), which will be initiated with once daily administration of the dose received TID in the CP. During MP, the Investigator is able to titrate the dose up or down in the range 2.5 g to 15 g body weight equivalent to maintain normokalaemia.

Long term Maintenance Phase (LTMP): For participants who, at the end of MP, are normokalaemic or hyperkalaemic without being on maximum dose, the MP is followed by the option to continue the study in a long term maintenance phase (LTMP) where the same titration regimen is used as in MP.

Data Monitoring Committee:

The iDMC will recommend on the opening of dose levels during the CP after reviewing all available data. Additionally, iDMC will recommend whether and when enrolment in the ages 0 to < 6 years cohorts will begin, and will also evaluate emerging safety data during all phases of the study.

Statistical methods: Objectives will be evaluated based on analysis populations corresponding to each study phase. Analysis sets are defined for each phase as the set of all participants who transitioned from previous phase and who received at least one dose of SZC during the phase. Primary assessments of the primary objectives, the probability to achieve and maintain normokalaemia when treated with SZC, will be based on point estimates together with 95% confidence intervals (CIs) from generalised linear models (repeated measures model for the MP). The secondary objective of change in S-K+ over time will be evaluated using a repeated measures linear model. Additional analyses, including analyses for other secondary objectives, will be done descriptively. In general, data will be analysed in the total analysis population, within each age cohort and, for the CP, within adult body weight equivalent dose-level, as appropriate. An interim read-out may be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent of the participant or legal representative, and informed assent from the participant (as appropriate)
2. Female or male from birth to < 18 years of age (for the study duration).
3. Participants (including those receiving a stable peritoneal dialysis regimen for a minimum of 2 months) requiring long-term treatment of hyperkalaemia (chronic hyperkalaemia) in the age cohort ≥ 2 years, and participants requiring either short- or long-term treatment for hyperkalaemia (acute and chronic hyperkalaemia) in the age cohort < 2 years.
4. Participants must meet the following criteria for hyperkalaemia: Please refer to the Table 6 in the protocol.
5. Using digital ECG, QT interval corrected by Bazett's method (QTcB) must meet the age-appropriate parameters at Screening: a. For participants aged 0 to ≤ 3 days after birth: < 450 ms b. For participants aged >3 days to < 12 years: < 440 ms c. For participants aged ≥ 12 to < 18 years: < 450 ms (male), < 460 ms (female) All QTcB values outside the reference values specified in the protocol should be manually re-measured and re-calculated, and if there is a difference in measurement between the automatic and manual ECG, the manual measurement should always be considered correct.
6. Ability to have repeated blood draws or effective venous catheterisation.
7. Females of childbearing potential (defined as a female with potential of becoming pregnant who has experienced her menarche) must have a negative pregnancy test within one day prior to the first dose of SZC on CP Study Day 1 and sexually active females of childbearing potential must be using 2 forms of medically acceptable contraception with at least one being a barrier method
8. Optional open-label, LTMP only:

   1. Provision of written informed consent of the participant or legal representative, and informed assent from the participant (as appropriate) to take part in the LTMP.
   2. Participants who are normokalaemic at the end of MP or hyperkalaemic and not on maximum dose.
   3. Participants who would benefit from long-term treatment for their hyperkalaemia, as judged by the Investigator.

Exclusion Criteria:

1. Neonates with a gestational age < 37 weeks at birth or a birth weight < 2500 g.
2. Term and preterm neonates with suspected conditions predisposing them to intestinal ischaemia (eg, perinatal hypoxia or sepsis).
3. Participants with pseudohyperkalaemia caused by excessive fist clenching to enable venepuncture, by haemolysed blood specimens, or by severe leukocytosis or thrombocytosis.
4. Participants with hyperkalaemia due to soft-tissue damage from crush injury or burns. 5. Participants with hyperkalaemia due to a secondary cause, such as dehydration, excessive use of K+ supplements, or drug use (eg, beta-adrenergic antagonists) and that would be more appropriately treated with other interventions (eg, fluid resuscitation, dose adjustments of medications).

6. Participants with transient iatrogenic hyperkalaemia (eg, due to treatment with tacrolimus).

7. Participants treated with lactulose, rifaximin (XIFAXAN™), or other nonabsorbed antibiotics for hyperammonaemia within the last 7 days.

8. Participants treated with CPS, sodium polystyrene sulfonate (eg, KAYEXALATE™), or patiromer within the last 4 days prior to first dose of study treatment.

9. Participants with a life expectancy of less than 3 months. 10. Participants who are known to have tested Human Immunodeficiency Virus (HIV) positive.

11. Presence of any condition which, in the opinion of the Investigator, places the participant at undue risk or potentially jeopardises the quality of the data to be generated. 12. Known hypersensitivity or previous anaphylaxis to SZC or to components thereof.

13. Participants with cardiac arrhythmias that require immediate treatment. 14. Participants with a family history of long QT syndrome. 15. Participants on haemodialysis. 16. Participants with a history of bowel obstruction. 17. Participants with severe gastrointestinal disorder or major gastrointestinal surgery (eg, large bowel resection).

18. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

19. Previous treatment with SZC. 20. Treatment with a drug or device within the last 30 days prior to first dose of study treatment that has not received regulatory approval at the time of study entry.

21. Previous enrolment in the present study. 22. Females who are pregnant, breastfeeding, or planning to become pregnant. 23. Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements. 24. If the participant has evidence of Coronavirus disease 2019 (COVID-19) within 2 weeks prior to enrolment (a positive COVID-19 test or suspicion of COVID-19 infection) the participant cannot be enrolled in the study.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2030-02-21 (Estimated); Study Completion 2030-02-21 (Estimated)

PRIMARY OUTCOMES:
Correction phase (CP) primary objective: To evaluate the ability to achieve normokalaemia during the CP when initiating treatment with SZC of different dose levels in children with hyperkalaemia | 3 days
  Normokalaemia achieved in the CP within 3 days (yes/no)
28-day Maintenance Phase (MP) primary objective: To evaluate the ability to maintain normokalaemia during the MP when continuing SZC treatment in children achieving normokalaemia | last two scheduled visits in the MP
  28-day MP primary endpoint: Serum potassium (S-K+) value within normokalaemia range (yes/no) at each of the last two scheduled visits in the MP

SECONDARY OUTCOMES:
All phases secondary objective: To evaluate the change in S-K+ in children treated with SZC | at each scheduled visit
  All phases secondary endpoint: S-K+ level at each scheduled visit
MP secondary objectives: To evaluate change in serum aldosterone levels in children treated with SZC during the MP | from baseline to Week 3 of the MP
  MP secondary endpoints: Change in serum aldosterone levels from baseline to Week 3 of the MP
MP Secondary objective: To evaluate change in serum electrolytes (including bicarbonate), spot urinary pH and urinary electrolytes levels in children treated with SZC during the MP | from baseline to week 3 of the MP
  Change in serum electrolytes (including bicarbonate), and spot urinary pH and urinary electrolytes from baseline to week 3 of the MP
Long-term MP (LTMP) secondary objectives: To evaluate the ability of maintaining normokalaemia in children treated with SZC during the LTMP | at each scheduled visit
  LTMP secondary endpoints: S-K+ value within normokalaemia range (yes/no) at each scheduled visit in the LTMP

OTHER OUTCOMES:
Safety objective: To evaluate the safety and tolerability of SZC in the 3 phases (CP, MP and LTMP) | Throughout the study, 27 weeks
  Adverse events/serious adverse events, Vital signs, Electrocardiogram, Clinical laboratory variables
Tertiary/Exploratory objective: To evaluate the acceptability and palatability of SZC through the study | At certain timepoints throughout the study
  Response categories in Study Medication Palatability Assessment questionnaires

CONTACTS AND LOCATIONS:
Locations (64):
- United States (14):
  - Research Site, Birmingham, Alabama
  - Research Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbia, South Carolina
  - Research Site, Morgantown, West Virginia
- Brazil (2):
  - Research Site, Campinas
  - Research Site, São Paulo
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Montreal, Quebec
- China (7):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Shanghai
- Germany (3):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Heidelberg
- India (3):
  - Research Site, Bhubaneshwar
  - Research Site, Gūrgaon
  - Research Site, New Delhi
- Japan (10):
  - Research Site, Bunkyō City
  - Research Site, Fuchu-shi
  - Research Site, Fukuoka
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Matsumoto-shi
  - Research Site, Nakagami-gun
  - Research Site, Saitama-Shi
  - Research Site, Sendai
  - Research Site, Shizuoka
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Research Site, Samara, Russia
- Spain (2):
  - Research Site, Esplugues de Llobregat
  - Research Site, Madrid
- Ukraine (6):
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Zaporizhzhia
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Hampshire
  - Research Site, Manchester
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home